CLINICAL TRIAL: NCT04272918
Title: Caregiver Support Model & Psycho-Education Program On Empowerment: Development and Validation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: City University of Hong Kong (Other)
Collaborators: Simon K.Y.Lee Foundation (Unknown)
Responsible Party: Principal Investigator, Dr. CHIU Yu Lung Marcus, Associate Professor, City University of Hong Kong
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: Carer Project
Record Dates: First submitted 2020-02-09; First posted 2020-02-17 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Caregiver Burnout; Case Management; Empowerment
Keywords: caregiver support; intensive case management; empowerment for caregivers
MeSH Terms: conditions — Caregiver Burden; Empowerment

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: For CSM, participants will not know their status (treatment vs control) and the existence of the other group. For PPE, there will be no masked information but exchange of information and cross discussion between two groups will be discouraged. For outcome assessment, a coordinator will be used and assessors will not know beforehand whether the case to assess is from treatment or control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- CSM condition (Experimental): Social Worker 1 of CSM conditions will work with caregivers according to the guidelines and template of the Care Support Model, including the formulation of the intervention plan based on CNA scores of different need domains, the use of the caregiver intervention plan template, service matching drawing reference from caregiver resource database, service formulation based on CNA scores of different strength domains, the use of the case monitoring template and guideline.
  Interventions: Behavioral: Caregiver Support Model
- Non-CSM condition (No Intervention): Social Worker 2 of the Control Group will not be notified of the CNA scores of his/her caregivers. The intervention plan, services assignment and case management of participants of the control group will be based on Social Worker 2's own judgement using the information shared by the caregivers, and the social worker's own observation.
- PP-E condition (Experimental): Experimental Group will be led a consultant who is an expert, with the help of a degree-holder social worker to facilitate capacity building, empowerment and long-term well-being. Measurement of outcome variables will be conducted before the start of the program, at the end of the program, and 3 months after the program ended.
  Interventions: Behavioral: Psycho-education Program
- Non PP-E condition (No Intervention): Measurement of outcome variables will be conducted at the same point of time as PP-E condition. There will be no treatment or intervention for the control group.

INTERVENTIONS:
Behavioral: Caregiver Support Model — Examine the effectiveness of the Caregiver Support Model (CSM) on improving caregivers' well-being.
  Arms: CSM condition
Behavioral: Psycho-education Program — Examine the effectiveness of the Psycho-education Program (PP-E) on capacity building, empowerment, and improving well-being.
  Arms: PP-E condition

SUMMARY:
This Project aims to provide social workers and relevant human service professionals with a comprehensive, scientific, and validated service model and suggest a sustainable support framework on the working process of helping and empowering family caregivers of frail elders, reducing caregiving distress, and enhancing caregivers' quality of life.

The proposed Project consists of two parts to be conducted in 1 year. The first part focuses on the development and validation of Caregiver Support Model (CSM) with a Randomized Controlled Trial (RCT) study. The second part develops and validates a psycho-education program on empowering family caregivers with another Randomized Controlled design. In the first year, the Project Team have (1) developed and designed different components of the Caregiver Support Model (CSM), including a comprehensive need assessment tool, personalized Caregiver Intervention Plan Guidelines and Template, and online database on caregiver services and community resources, (2) designed a five-session psycho-education program on empowerment. The Caregiver Needs Assessment (CNA) tool was also pilot-tested with 320 community caregivers. Results from the survey, together with the systematic review on caregiver support, will form the backbone of the later CNA implementation. The working model will be validated using RCT design with 400 family caregivers recruited through 4 collaborating NGOs. At the same time, a psycho-education program on empowerment will be developed and validated using RCT design with another 190 caregivers.

DETAILED DESCRIPTION:
Participants of CSM will be randomly assigned to CSM intervention and non-CSM intervention which is the usual practice of case handling by centre staff. Randomization will be based on centres to prevent exchange of information between the two groups, and thus causing contamination. Outcome data will be measured at 3 time-intervals: case intake, 3-month, and 6-month.

Participants of the psychoeducation program on empowerment (PPE) will be randomly assigned to the program group and the non-program group. For the former a 5-session psychoeducation program will be administered. For both groups, outcome measures will be collected at pre, post, and 3-month after post test.

ELIGIBILITY:
CSM Inclusion Criteria:

* Primary family caregivers aged 21 or above;
* Have not received major/ intensive services in the past three months;
* Providing care for elderly aged 60 or older;
* Care recipient has at least one difficulty in activities of daily living or instrumental activities of daily living that needs help from the caregiver (scored 3 or higher on at least one of the items in the ADL/IADL Checklist).

PPE Inclusion Criteria:

* Primary family caregivers aged 21 or above;
* Family caregiving in stable situation or care recipient passed away within 2 years;
* Have not received systematic psychoeducation in the past three months.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 590 (Estimated)
Dates: Start 2020-02-15 (Estimated); Primary Completion 2020-12-30 (Estimated); Study Completion 2021-08-15 (Estimated)

PRIMARY OUTCOMES:
Change of score in Zarit Burden Interview (Zarit, Reever, Bach-Peterson, 1980) | CSM: Change between baseline, 3 months and 6 months
  Zarit Burden Interview is a 12-item scale, and each item is scored 1 to 5 (1 = never; 5 = Always). It measures subjective burden among caregiver of adults with dementia, including functional/behavioral impairments and home care situation. Items are worded to focus on the affective response of the caregiver.
Change of score in WHO-5 (Topp et al. 2015) | CSM: Change between baseline, 3 months and 6 months
  The WHO-5 is a short questionnaire consisting of 5 simple and non-invasive questions, which access 5 aspects of subjective well-being of the respondents Each of the 5 items is scored from 5 (all of the time) to 0 (none of the time).
Change of score in Meaning in caregiving (Yen et al., 2009) | PPE: Change between Baseline, 1 month and 3 months
  Meaning in caregiving was measured via the 12-item Meaning in Caregiving Scale developed by Ciuliano et al. (1990), translated by Yen et al., 2009. The instrument used a 5-point Likert scale: 1 (Strongly Disagree) to 5 (Strongly Agree).
Change of score in Attitudes towards helping others (Webb, Green & Brashear，2000) | PPE: Change between Baseline, 1 month and 3 months
  Attitude toward helping others (AHO) is a 4-item measurement developed by Webb, Green and Brashear (2000) to measuring one's tendency to help or assist other people. Respondents answer each item using a 5-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree).
Change of score in Revised scale for caregiving self-efficacy (Steffen et al., 2002) | PPE: Change between Baseline, 1 month and 3 months
  The RSCSE is a 15-item measurement which can assesses caregivers' confidence in responding to three domains of caregiving: obtaining respite, managing disruptive behaviors, and controlling upsetting thoughts. The scale is scored from 0 (cannot do at all) to 10 (certain can do).
Change of score in Family Empowerment Scale (Koren, DeChillo and Friesen, 1992) | PPE: Change between Baseline, 1 month and 3 months
  The Family Empowerment Scale is a 34-item questionnaire developed by Koren, DeChillo and Friesen (1992) for assessing the 3 aspects of empowerment in family: family, service and community. A 5-point scale is used (1 = not at all; 5 = very true).
Change of score in 5-level EQ-5D (EQ-5D-5L; EuroQol Group, 2009) | CSM: Change between baseline, 3 months and 6 months
  The 5-level EQ-5D version (EQ-5D-5L) was introduced by the EuroQol Group (2009), assessing five dimensions including mobility, self-care,, usual activities, pain/discomfort and anxiety/depression on a 5-point scale, ranging from 1 to 5 (1 = no problem at all; 5 = extremely worse condition)
Change of score in General Health Questionnaire-12 (Goldberg & Williams, 1988) | CSM: Change between baseline, 3 months and 6 months
  The General Health Questionnaire-12 is a shortened version of the General Health Questionnaire scored on a 4-point scale, developed by Goldberg and Williams (1998), designed to measure the risk of developing psychiatric disorders and assess general well-being of a person.
Change of score in 7-item Peace of Mind Scale (Lee et al., 2013) | CSM: Change between baseline, 3 months and 6 months
  The Peace of Mind Scale consist of 7 items, measuring one's internal state of peacefulness and harmony among Chinese culture. It is scored 1 to 5 (1 = never; 5 = always)

CONTACTS AND LOCATIONS:
Overall Officials: Tit-wing LO, Study Director — City University of Hong Kong; Kin-Kit (Ben) LI, Study Director — City University of Hong Kong; Yuen Lan Dannii YEUNG, Study Director — City University of Hong Kong
Locations (1):
- City University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zarit SH, Reever KE, Bach-Peterson J. Relatives of the impaired elderly: correlates of feelings of burden. Gerontologist. 1980 Dec;20(6):649-55. doi: 10.1093/geront/20.6.649. No abstract available. PMID 7203086
- [Background] Topp CW, Ostergaard SD, Sondergaard S, Bech P. The WHO-5 Well-Being Index: a systematic review of the literature. Psychother Psychosom. 2015;84(3):167-76. doi: 10.1159/000376585. Epub 2015 Mar 28. PMID 25831962
- [Background] Yen WJ, Huang XY, Ma WF, Lee S, Lee CH. A Chinese version of the Meaning in Caregiving Scale: an assessment of its reliability and validity. Perspect Psychiatr Care. 2009 Apr;45(2):140-50. doi: 10.1111/j.1744-6163.2009.00214.x. PMID 19366424
- [Background] Webb, D. J., Green, C. L., & Brashear, T. G. Development and validation of scales to measure attitudes influencing monetary donations to charitable organizations. Journal of the academy of marketing science, 28(2), 299-309, 2000
- [Background] Steffen AM, Gallagher-Thompson D, Arenella KM, Au A, Cheng ST, Crespo M, Cristancho-Lacroix V, Lopez J, Losada-Baltar A, Marquez-Gonzalez M, Nogales-Gonzalez C, Romero-Moreno R. Validating the Revised Scale for Caregiving Self-Efficacy: A Cross-National Review. Gerontologist. 2019 Jul 16;59(4):e325-e342. doi: 10.1093/geront/gny004. PMID 29546334
- [Background] Koren, P. E., DeChillo, N., & Friesen, B. J. Measuring empowerment in families whose children have emotional disabilities: a brief questionnaire. Rehabilitation psychology, 37(4), 305, 1992.
- [Background] Lou VW, Lau BH, Cheung KS. Positive aspects of caregiving (PAC): scale validation among Chinese dementia caregivers (CG). Arch Gerontol Geriatr. 2015 Mar-Apr;60(2):299-306. doi: 10.1016/j.archger.2014.10.019. Epub 2014 Nov 7. PMID 25488014
- [Background] Goldberg, D., & Williams, P. General health questionnaire (GHQ). Swindon, Wiltshire, UK: nferNelson, 2000.
- [Background] Lee, Y. C., Lin, Y. C., Huang, C. L., & Fredrickson, B. L. The construct and measurement of peace of mind. Journal of Happiness studies, 14(2), 571-590, 2013